CLINICAL TRIAL: NCT03922269
Title: Trans People Living With HIV Throughout Europe
Acronym: TIME
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: C&W19/003
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Gender Identity; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender individual with a diagnosis of HIV: The participant self-identifies as transgender and/or has a current gender identity which differs from gender assigned at birth, is 18 years old or above, has a diagnosis of HIV infection and has been prescribed antiretroviral therapy.

SUMMARY:
The project will study a European cohort of individuals identifying themselves as transgender or non-binary and living with HIV.

The study will collect both qualitative data on this cohort and clinical data over an 18 month period. The study will investigate the success of HIV treatment for this cohort through the primary outcome measure of HIV viral load recorded in routine blood tests.

The results from this study will assist in informing future HIV treatment guidelines on the monitoring of HIV infection in transgender and non-binary individuals and assisting in the design of future interventional studies within this population.

DETAILED DESCRIPTION:
The TIME Study is a multi-centre cohort study, combined with a cross-sectional survey.The study will comprise recording clinical data from up to three visits over an 18-month period. The study visits will happen at the same time of routine clinical care, and all clinical data will be collected in the study database. At the screening/baseline study visit (following written consent), a survey will be administered to all study participants. The overall recruitment target is 200 participants.

The primary aim is to assess the rate of virological response to antiretroviral therapy in transgender and non-binary (gender diverse) people living with HIV (TPLWH) in Europe. It's secondary outcomes are:

* To explore demographics, risk behaviours and community needs
* To explore the barriers and facilitators to adherence to cART
* To report TPLWH experiences with regard to:

  * Stigma
  * Quality of life
  * Prevalence of opportunistic infections
* To record data on:

  * Retention into care
  * Clinical characteristics (e.g. drug toxicity, BMD results, hormone intake, drug interactions between hormones and antiretrovirals, cardiovascular risk, etc.)
* Implement and analyse a trans-inclusive method of gender identity data collection, in order to provide comprehensive demographic information that is acceptable at the community-level and includes a diverse spectrum of trans/non-binary genders across all study sites. People living with HIV (PLWH) who refer to themselves as transgender and non-binary (and all gender diverse people).

ELIGIBILITY:
Inclusion Criteria:

* Participant self-identifies as transgender and/or has a current gender identity which differs from gender assigned at birth (includes all gender diverse people)
* Age > 18 years
* HIV infection diagnosis at any time before study consent
* Having been prescribed antiretroviral therapy at any time (including people for who antiretroviral therapy initiation is planned after study enrolment)
* Willing to sign an informed consent and take part in the study

Exclusion Criteria:

* Age < 18 years
* Unable to take part in the study according to the Investigator opinion (example: unable to understand the study information leaflet, unable to provide written consent, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant self-identifies as transgender and/or has a current gender identity which differs from gender assigned at birth (includes all gender diverse people).
Study Population: Participant self-identifies as transgender and/or has a current gender identity which differs from gender assigned at birth (includes all gender diverse people) They must be 18 years old or above, have a diagnosis of HIV and have been prescribed antiretroviral therapy at any time.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Rate of virological response to antiretroviral therapy | 18 months
  Proportion of cohort achieving viral suppression as measured in viral load serum assays.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD, PhD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (4):
- Servizio Sanitario Nazionale Regione Piemonte Azienda Sanitaria Locale "Citta di Torino" Department of Medical Sciences, University of Turin, Torino, Italy
- United Kingdom (3):
  - Chelsea and Westminster Hospital, London, Greater London
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Elton John Centre, Brighton and Sussex University Hospitals, Brighton, Sussex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baral SD, Poteat T, Stromdahl S, Wirtz AL, Guadamuz TE, Beyrer C. Worldwide burden of HIV in transgender women: a systematic review and meta-analysis. Lancet Infect Dis. 2013 Mar;13(3):214-22. doi: 10.1016/S1473-3099(12)70315-8. Epub 2012 Dec 21. PMID 23260128
- [Background] Suchak et al. Highly invisible, highly infectious and high risk: the hidden problem of trans people living with HIV. 23rd Annual Conference of the British HIV Association (BHIVA), 2017. Liverpool, UK.
- [Background] Santos GM, Wilson EC, Rapues J, Macias O, Packer T, Raymond HF. HIV treatment cascade among transgender women in a San Francisco respondent driven sampling study. Sex Transm Infect. 2014 Aug;90(5):430-3. doi: 10.1136/sextrans-2013-051342. Epub 2014 Apr 8. PMID 24714446
- [Background] Hibbert M, Wolton A, Crenna-Jennings W, Benton L, Kirwan P, Lut I, Okala S, Ross M, Furegato M, Nambiar K, Douglas N, Roche J, Jeffries J, Reeves I, Nelson M, Weerawardhana C, Jamal Z, Hudson A, Delpech V. Experiences of stigma and discrimination in social and healthcare settings among trans people living with HIV in the UK. AIDS Care. 2018 Jul;30(7):836-843. doi: 10.1080/09540121.2018.1436687. Epub 2018 Feb 6. PMID 29409344
- [Background] Herbst JH, Jacobs ED, Finlayson TJ, McKleroy VS, Neumann MS, Crepaz N; HIV/AIDS Prevention Research Synthesis Team. Estimating HIV prevalence and risk behaviors of transgender persons in the United States: a systematic review. AIDS Behav. 2008 Jan;12(1):1-17. doi: 10.1007/s10461-007-9299-3. Epub 2007 Aug 13. PMID 17694429
- See also: HIV/AIDS surveillance in Europe 2018 - 2017 data — https://ecdc.europa.eu
- See also: UNAIDS — http://www.unaids.org
- See also: WHO policy brief - Transgender people and HIV — http://www.who.int